CLINICAL TRIAL: NCT04571866
Title: The Effect of Dietary Fiber-enriched Bread on Gastric Emptying and Postprandial Glucose Levels
Brief Title: Gastric Emptying After Bread Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Jutta Dierkes, Professor, University of Bergen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 120533
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Gastric Emptying
Keywords: Gastric emptying; Carbohydrate; Bread consumption; Beta-glucan; Metabolic response

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-glucan bread (Experimental): Participants will receive a standardised meal consisting of beta-glucan-enriched bread (in an amount corresponding to 25 g of available dietary carbohydrates) and water (250 ml). The bread is produced by NOFIMA AS, one of the collaborating parties. The participants will be asked to spend approximately 10 minutes consuming the standardised meal.
  Interventions: Other: Beta-glucan bread
- Control bread (Sham Comparator): Participants will receive a standardised meal consisting of a wheat bread with no additives (in an amount corresponding to 25 g of available dietary carbohydrates) and water (250 ml). The bread is produced by NOFIMA AS, one of the collaborating parties. The participant will be asked to spend approximately 10 minutes consuming the standardised meal.
  Interventions: Other: Beta-glucan bread

INTERVENTIONS:
Other: Beta-glucan bread — Beta-glucan is a dietary fiber with beneficial health effects, both on cholesterol levels and potentially blood glucose levels.

SUMMARY:
The rate of gastric emptying is proposed to be one of the major determinants of postprandial glycemia. A slower gastric emptying will thus result in a less pronounced rise in blood glucose, which is especially desirable in diabetes care as it will highly influence the overall glycemic control. The present study aims to investigate the rate of gastric emptying and postprandial blood glucose levels in response to the intake of bread with different dietary fiber-content. Though bread is one of the major sources of dietary carbohydrates in Central- and Northern Europe, the mechanism and the metabolic effects of bread consumption, however, is investigated in a limited number of studies.

DETAILED DESCRIPTION:
The rate of gastric emptying is related to small intestinal motility and absorption of carbohydrates, and it is one of the major determinants of postprandial glycemia. A slower rate of gastric emptying will thus result in a less pronounced rise in blood glucose. Especially in diabetes care, reduced gastric emptying is desirable because of its effect on the rise of postprandial blood glucose, which again highly influences the overall glycemic control.

Bread is one of the most eaten food items in Central- and Northern Europe, being one of the major sources of dietary carbohydrate intake. In addition, bread often contains a diverse range of dietary fiber. The effect on gastric emptying and the amount of dietary carbohydrates absorbed in the small intestine depends on the overall meal composition, the degree of processing, and the type of dietary fiber, e.g., viscous or non-viscous. The oat-derived dietary fiber beta-glucan may have favorable properties in this regard as adding beta-glucan to a meal has been shown to slow down the rate of gastric emptying. However, studies investigating the effect of beta-glucan on gastric emptying are scarce.

For assessment of gastric emptying, scintigraphy is seen as the "gold standard" as the method readily can discriminate between gastric emptying and absorption of glucose in the small intestine. However, this method is not often used due to its invasive nature and radiation. High-resolution real-time ultrasonography is now the most preferred method and regarded as a new "gold standard", proving good inter- and intra-observer agreement. Compared to scintigraphy, ultrasound is a safe and non-invasive procedure widely available in clinical settings.

Objectives

To establish whether a wheat bread with an optimized content of beta-glucan has a different effect on gastric emptying, satiety, and postprandial glycemia compared to control bread.

Study procedures

Recruitment

Healthy adults (age range 18 to 40 years) with normal to overweight body mass index (BMI: 18.5-30 kg/m2) and no gastrointestinal diseases or other issues that can affect gastric motility, are eligible and will be asked to participate. Health status will be briefly checked during a screening examination.

Participants will be recruited through flyers, announcements, and advertisements in social media, such as Facebook. The eligibility of participants will be addressed during a screening visit. Participants will answer questionnaires including questions on general health status, lifestyle habits, current medications, allergies, and gastrointestinal symptoms (using the ROMA-IV questionnaire).

Study design: randomized cross-over design

The study will be conducted at the Research Unit for Health Surveys, University of Bergen, on non-consecutive days, with at least 3 days (wash-out period) in between two study days. Participants will consume bread with either beta-glucan or no additive at a quantity of 25 g available carbohydrates within 10 minutes together with 250 ml water. Gastric emptying will then be measured by ultrasound during the next 2 hours in 15 minute-intervals the first hour, and then every 30th minute (15, 30, 45, 60, 90, and 120 minutes). Blood samples will be taken for measurement of postprandial glucose and satiety hormones, and the participants will fill in a Visual Analogue Scale (VAS) for satiety. Blood pressure, body weight, waist circumference, and height will be measured during the study visit. The participants must be fasting for at least 12 hours (overnight, usually from 8 pm the evening before the study visit).

Study bread will be blinded to both the investigators and the participants, although it cannot be excluded that participants may recognize the type of bread. Consumption of bread occurs in a randomized order, according to a randomization scheme.

Gastric emptying by ultrasound

Measurement: The participant is to be placed in a standardized sitting position. The cross-sectional area of the antrum of the stomach will be measured using 2D ultrasonography. The outer profile of the antrum will be measured using a built-in caliper and a calculation program available in the ultrasound apparatus. The gastric antrum, the mesenteric vein, and the aorta have to be visualized in this section. A minimal amount of force must be applied during each reading to prevent compression of the antrum. The measurement will be performed when the participants are suspending their breathing in expiration, between antral contractions. The average of the two measurements will be used.

The antral area will be measured at the fasting state (baseline), immediately following bread and water intake, and during the next 2 hours at regular intervals.

Blood glucose and satiety hormones

The effect of gastric emptying on postprandial blood glucose will be measured by collecting venous and capillary blood samples. Venous blood samples, sampled via a catheter inserted into an arm vein, will be collected at baseline, and 15, 30, 45, 60, 90, and 120 minutes after the participant starts to ingest the test meal. In addition, the venous blood samples will be used for the determination of insulin, Glucagon-like peptide-1 (GLP-1), peptide YY (PYY), ghrelin, and leptin. The capillary blood samples, collected at the same time intervals as the venous blood samples, will be used to measure postprandial blood glucose levels.

Satiety

The participants will be asked to report satiety sensations by filling in a VAS at baseline, and 15, 30, 45, 60, 90, and 120 minutes after consumption of the standardized meals, without having the previous scale available.

Statistics

The primary outcome variable is the difference in gastric emptying (antral area, cm2) at different time points and the calculated area under the curve for the entire study duration. The comparison of the antral area following the different bread-options will be done at each time point using a Tukey's multiple comparisons test. Each subject serves as her/his control when comparing antral areas at different time points.

Secondary outcomes are the postprandial blood glucose concentrations at different time points, subjectively reported satiety, insulin, and satiety hormones at different time points.

Ethics

Participants will be provided with written and oral information about the study. Before inclusion, the participants have to sign a consent form. The participants can withdraw from the study at any time without explanation. The study will be performed following the Declaration of Helsinki.

Overall, participation in the study implies very little risk. Some discomfort may occur when drawing blood and bruising can occur. However, blood sample collection will be performed by authorized personnel in a standardized matter. Participants will be covered by the Patient Injury Act.

All study procedures will be conducted in accordance with Good Clinical Practice. All study procedures will be described in standard operating procedures (SOPs).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-40 years
* BMI: 18.5-30 kg/m2
* Healthy

Exclusion Criteria:

* Celiac disease, non-celiac gluten sensitivity or wheat allergy and intolerance
* Use of medication that can affect gastric emptying
* Gastroparesis
* Gastrointestinal diseases
* Gastrointestinal surgery including bariatric surgery
* Chronic alcohol abuse
* Current smoker
* Pregnant or lactating women
* Diabetes mellitus type 1 and 2
* Anorexia nervosa or bulimia nervosa

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Difference in gastric emptying (antral area, cm2) ) | 2 hours
  Differences in antral area (cm2) at different time points after ingestion of standardised meals. The antral area is measured by real-time ultrasonography.

SECONDARY OUTCOMES:
Satiety hormones | 2 hours
  Differences in the concentration of GLP-1, PYY -, leptin and ghrelin
Subjective satiety | 2 hours
  Differences in the reporting of satiety sensation using a Visual analog scale (VAS; scale 0-10, 0=extremely hungry/not hungry at all, 10= extremely full/extremely hungry )
Postprandial blood glucose | 2 hours
  Differences in postprandial blood glucose measured at different time points
Insulin | 2 hours
  Differences in postprandial insulin measured at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Dierkes, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Derived] Revheim I, Ballance S, Standal AF, Rieder A, Dierkes J, Buyken AE, Gilja OH, Hausken T, Rosendahl-Riise H. The acute effect of a beta-glucan-enriched oat bread on gastric emptying, GLP-1 response, and postprandial glycaemia and insulinemia: a randomised crossover trial in healthy adults. Nutr Metab (Lond). 2024 Mar 18;21(1):13. doi: 10.1186/s12986-024-00789-w. PMID 38500209